CLINICAL TRIAL: NCT06485349
Title: Olive Leaf Extract Effects on Meta-inflammation and Anxiety Symptoms in Women With Excess Weight
Brief Title: Olive Leaf Extract, Meta-inflammation, Anxiety, and Excess Weight
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Ma. Sonia Luquín de Anda, Principal Investigator, Head of Neuroscience Department, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-11
Record Dates: First submitted 2024-06-14; First posted 2024-07-03 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Women; Excess Weight; Anxiety Disorders
Keywords: Olive leaf extract; Women; Meta-inflammation; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — olive leaf extract; oleuropein

STUDY DESIGN:
Intervention Model Description: Excess-weight women with mild anxiety symptomatology will be assigned in a control double-blind and randomized manner to one of two groups: olive leaf extract (OLE) (n=35) 750 mg 20% oleuropein or placebo (n=35). Participants would have sessions biweekly:
  1. (Day 0, 30, 60, and 90): Anxious symptomatology, weight, height, body fat, and muscle percentage (blood extraction at day 0 and day 90).
  2. (Day 15, 45, 75): Adherence, 24-hour recall, and Food frequency questionnaire (FFQ).
  Supplementation starts at day 0 and ends at day 89. Anxious symptomatology is evaluated, monthly, alternatively with the Hamilton Anxiety Scale (HAS) and Beck Anxiety Inventory (BAI). Adherence will be verified every 15 days as well as a 24-hour dietary recall and FFQ. ELISA assays will be used for TNF-α, IL-6, Cortisol, and leptin quantifications. It will be performed with 12h overnight fasting, in the morning; and lipid profile and glycosylated hemoglobin will be measured through biochemical tests.
Who Masked: Participant, Investigator
Masking Description: double-blinded control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Olive Leaf Extract (OLE) Nutricost ® 750mg 20% oleuropein with 250ml of water.
  Interventions: Dietary Supplement: Olive Leaf Extract (OLE)
- Placebo (Placebo Comparator): 100mg cellulose with 250ml of water.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Olive Leaf Extract (OLE) — Daily dose of 750mg OLE consumed with water after breakfast without any modification of their dietary patterns for 90 days.
  Other Names: Olive leaf extract Nutricost ® 750mg 20% oleuropein
  Arms: Experimental
Other: Placebo — 100mg microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Excess Weight is accompanied by a process that produces a low-grade inflammation state, called meta-inflammation. Anxiety is also associated with inflammation. Inflammation is closely related to oxidative stress. Both processes help perpetuate each other. Olive Leaf Extract (OLE) is known for having anti-inflammatory and antioxidant effects; by this means, its anxiolytic effect has been proved in animal models. The purpose of this investigation is to evaluate the anti-inflammatory and anxiolytic effects associated with the supplementation of OLE at a daily dose of 750mg (20% oleuropein) for 3 months.

DETAILED DESCRIPTION:
A randomized double-blind placebo clinical trial is proposed. Study groups will be comprised of women living with excessive weight from the Guadalajara Metropolitan Area who meet the following criteria: age ≥18- ≤40 years, body mass index (BMI) ≥25- ≤40 kg/m^2, blood pressure ≤ 129 mmHg systolic and ≤80 diastolic; anxiety symptomatology score 6 to 14 (mild) according to Hamilton Anxiety Scale (HAS).

70 women at the University Center for Health Sciences (CUCS) from Universidad de Guadalajara who meet inclusion criteria will be invited to participate. Two groups will be randomly formed consisting of 35 women with excessive weight and anxious symptoms each (by the BMI and HAS score, respectively); 35 will receive cellulose (100 mg) as a placebo, and the other 35, 750 mg/day of Olive Leaf Extract (OLE) orally, daily, for 90 days. Participants would be instructed to consume it after breakfast without modifying their eating patterns.

Anxious symptomatology will be measured by HAS and Beck Anxiety Inventory (BAI), alternately, every 30 days for 90 days; at the beginning, it would be HAS, after 30 days, investigators will apply BAI, then, after the next thirty days HAS (day 60) and, finally, will end the study applying BAI (day 90). Alternation of these tests is done to avoid bias in patients that allows them to recognize answers to obtain better scores.

Treatment adherence will be reviewed on a biweekly basis. At the same time, biweekly, participants will have to fill out a nutritional 24-hour food recall and a food frequency questionnaire and will also be asked if it is their desire to keep participating or not in the investigation.

To evaluate meta-inflammation, levels of leptin, IL-6, TNF-α, and cortisol in serum will be quantified using the ELISA technique. This will be done by doing a blood extraction at the beginning and another one at the end of the study (day 90). These two extractions will also be used to measure the patient's lipid profile (LDL cholesterol; LDL-c, total cholesterol; TC, triglycerides; TG and HDL-cholesterol; HDL-c) and glycosylated hemoglobin.

At the beginning of the study, investigators will apply a nutritional clinic history that contains information on eating habits (24-hour recall and food frequency), clinical history, and family health history. Anthropometric parameters such as weight, height, age, and BMI will be recorded; also, the percentage of body fat and muscle through bioimpedance. Height will be measured with a stadiometer. Weight and components associated with excessive weight such as percentage of body fat and muscle will be recorded monthly using an Omron® HBF-514C bioimpedance scale.

ELIGIBILITY:
Inclusion Criteria:

* Females.
* Residing in Guadalajara Metropolitan Area (GMA).
* Initial age ≥18-≤ 40 years
* Initial Body Mass Index (BMI) ≥25-≤40 kg/m^2
* Blood pressure: ≤129mmHg systolic and ≤80 diastolic.
* Anxious symptomatology score 6 to 14 (mild) through the Hamilton Anxiety Scale (HAS).

Exclusion Criteria:

* Use of psychoactive drugs, suffering from major psychiatric disorders (depression, attention deficit hyperactivity disorder, bipolar disorder, eating disorders), pregnancy, breastfeeding, hypotension, alcohol use disorder (AUD).
* Suffer from liver, kidney, or thyroid disease or cancer.
* Olive allergy.
* Consume any medication that influences weight
* Consume some other type of food supplement from organic origin.
* Less than 70% adherence frequency to the consumption of the extract/placebo.
* Getting pregnant during the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in TNF-α concentration | Baseline, day 0, pre-supplementation, on an empty stomach, and day 90 (on an empty stomach, 24 hours after the last supplement/placebo intake).
  Measured by ELISA assay (Enzyme-Linked ImmunoSorbent Assay) according to the manufacturer's recommendations. The kit is a Human TNF-α ELISA kit; measured in pg/mL.
Change in IL-6 concentration | Baseline, day 0, pre-supplementation, on an empty stomach, and day 90 (on an empty stomach, 24 hours after the last supplement/placebo intake).
  Measured by ELISA assay (Enzyme-Linked ImmunoSorbent Assay) according to the manufacturer's recommendations. The kit is a Human IL-6 ELISA kit; measured in pg/mL
Change in leptine concentration | Baseline, day 0, pre-supplementation, on an empty stomach, and day 90 (on an empty stomach, 24 hours after the last supplement/placebo intake).
  Measured by ELISA assay (Enzyme-Linked ImmunoSorbent Assay) according to the manufacturer's recommendations. The kit is a Human leptin ELISA kit; measured in pg/mL
Change in cortisol concentration | Baseline, day 0, pre-supplementation, on an empty stomach, and day 90 (on an empty stomach, 24 hours after the last supplement/placebo intake).
  Measured by ELISA assay (Enzyme-Linked ImmunoSorbent Assay) according to the manufacturer's recommendations. The kit is a Human cortisol ELISA kit; measured in pg/mL.
Change in Anxiety symptomatology scored by Hamilton Anxiety Scale (HAS) | From baseline, day 0, pre-supplementation, up to day 60, during supplementation. It will be applied bimonthly, twice in total.
  Measured in accordance to the next score: 0-5, absence of anxiety; 6-14, mild anxiety; ≥15, moderate/severe anxiety, on an alternately, monthly, basis; in the morning in a peaceful controlled environment.
Change in Anxiety symptomatology scored by Beck Anxiety Index (BAI) | Its first application will be on day 30, during supplementation, up to day 90 (24 hours after the last supplement/placebo intake). It will be applied bimonthly, twice in total.
  Measured in accordance to the next score: 0-5, absence of anxiety; 6-15, mild anxiety; 16-30, moderate anxiety; 31-63 severe anxiety, on an alternately, monthly, basis; in the morning in a peaceful controlled environment.

SECONDARY OUTCOMES:
Change in weight | From baseline, day 0, pre-supplementation. Then, during supplementation it will be measured monthly, meaning day 30, day 60 up to day 90 (24 hours after the last supplement/placebo intake).
  In kilograms (kg). Measured every month, in the morning, lightly clothed, with an Omron® HBF-514C bioimpedance scale in a peaceful controlled environment.
Change in body fat percentage | From baseline, day 0, pre-supplementation. Then, during supplementation it will be measured monthly, meaning day 30, day 60 up to day 90 (24 hours after the last supplement/placebo intake).
  Expressed in percentage (%). Measured every month, in the morning, lightly clothed, with an Omron® HBF-514C bioimpedance scale in a peaceful controlled environment.
Change in body muscle percentage | From baseline, day 0, pre-supplementation. Then, during supplementation it will be measured monthly, meaning day 30, day 60 up to day 90 (24 hours after the last supplement/placebo intake).
  Expressed in percentage (%). Measured every month, in the morning, lightly clothed, with an Omron® HBF-514C bioimpedance scale in a peaceful controlled environment.
Change in lipid profile | Baseline, day 0, pre-supplementation, on an empty stomach, and day 90 (on an empty stomach, 24 hours after the last supplement/placebo intake).
  Total cholesterol, triglycerides, high-density lipoprotein, low-density lipoprotein: Blood serum would be taken from the participants after an overnight fast of 12 h; lipid profiles (triglycerides, total cholesterol, HDL-C, and LDL-C) would be determined using a piece of semi-automated equipment (Mindray-BS-240 Clinical Chemistry Analyzer, Shenzhen, China) and colorimetric enzymatic assays (BioSystems® kits, Barcelona, Spain). Measured in mg/dl.
Change in glycosylated hemoglobin | Baseline, day 0, pre-supplementation, on an empty stomach, and day 90 (on an empty stomach, 24 hours after the last supplement/placebo intake).
  Blood serum would be taken from the participants after an overnight fast of 12 h; glycosylated hemoglobin would be determined using a piece of semi-automated equipment (Mindray-BS-240 Clinical Chemistry Analyzer, Shenzhen, China) and colorimetric enzymatic assays (BioSystems® kits, Barcelona, Spain). Measured in percentage (%).
24 hour dietary intake recall | Its first application will be on day 15, during supplementation. Then, it will be applied on a biweekly basis, meaning day 30, day 45, day 60, day 75 up to day 90 (24 hours after the last supplement/placebo intake).
  Taken on a biweekly basis to analyze the dietary intake consumed the previous day and measure their approximate caloric intake and macronutrient relationship with the Mexican Food Equivalent System.
Food Frequency Questionnaire | Its first application will be on day 15, during supplementation. Then, it will be applied on a biweekly basis, meaning day 30, day 45, day 60, day 75 up to day 90 (24 hours after the last supplement/placebo intake).
  Taken on a biweekly basis to analyze their food consumption according to their group classification.
Change in BMI | From baseline, day 0, pre-supplementation. Then, during supplementation it will be measured monthly, meaning day 30, day 60 up to day 90 (24 hours after the last supplement/placebo intake).
  Weight and height will be combined to report BMI in kg/m^2 and it will be measured every month according to their actual weight-height relation.

CONTACTS AND LOCATIONS:
Overall Officials: Ma. Sonia Luquin, Ph.D, Principal Investigator — University of Guadalajara
Locations (1):
- Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available. It will only be shared the data that underlie the results reported in this article, after deidentification. The study protocol, statistical analysis plan, and informed consent form are already in the document attached to this registry.
  Data will be available beginning 3 months and ending 2 years after article publication.
  It will be shared with anyone who provides a methodologically sound proposal, to achieve its aims. The proposal should be directed to sonia.luquin@academicos.udg.mx or to mario.hernandez6110@alumnos.udg.mx. To gain access, data requestors will need to sign a data access agreement.
  Data will be available to the requestors at this link: https://drive.google.com/drive/folders/1tL75USV4bsrOAvb5A-7-H3CcOowq-T1V?usp=drive_link
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available approximately 3 months after publication and it will end its availability after 2 years of it. After that period, if requested, data should be asked to sonia.luquin@academicos.udg.mx or to mario.hernandez6110@alumnos.udg.mx, subject to availability.
Access Criteria: The information will be available for research purposes to colleagues interested in the results of this study and whose information is useful to expand associated knowledge.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT06485349/Prot_SAP_ICF_000.pdf